CLINICAL TRIAL: NCT01708200
Title: A Comparison of the Effectiveness of Two Types of Cognitive Training Interventions Administered to Individuals With a Diagnosis of a Mental Health Condition.
Brief Title: A Comparison of the Effectiveness of Two Types of Memory Training Programs in People With a Diagnosis of Mental Illness.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Bruno Losier, Clinical Neuropsychologist, St. Joseph's Healthcare Hamilton
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: R.P. #12-3749; SJHH (Other: St. Joseph Healthcare Hamilton)
Record Dates: First submitted 2012-10-10; First posted 2012-10-16 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Memory Impairment
Keywords: Memory; Intervention; Computerized; Psychoeducational; Mental Illness
MeSH Terms: conditions — Memory Disorders; Mental Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Memory Intervention (Experimental): Two types of memory protocols (psychoeducational vs computerized) will be compared in a population of individuals with mental illness.
  Interventions: Other: Memory Intervention

INTERVENTIONS:
Other: Memory Intervention — A comparison of two type of memory intervention protocols; a psychoeducational/intervention protocol versus a computerized memory protocol in a population of individuals with mental illness.

SUMMARY:
This study will compare the effectiveness of a psychoeducational memory program versus a computerized memory program in individuals with mental illness. Although improvements are expected with both form of interventions, we do not know which will provide maximal benefit in this population.

DETAILED DESCRIPTION:
The aim of the current study is to compare two memory strategies, a top-down (i.e., educational and interventional)protocol vs. a bottom-up (computerized)protocol, in a population of individuals diagnosed with mental illness. Performance on ecologically validated memory tasks will be measured before and after each intervention protocol. Improvements are expected following each protocol. However, there is no evidence available to support added benefits from one protocol over another. As such, the current study will endeavour to contrast the two intervention types (top-down vs. bottom-up) to determine which, if any, provides maximal benefit.

ELIGIBILITY:
Inclusion Criteria:

* Memory impairment equivalent to 1.5 std. dev. below average for age
* Speak and read English fluently

Exclusion Criteria:

* Older than 65 years of age
* Significant visual impairment (e.g., cataracts, macular degeneration)
* Motor impairment (e.g., hemiplegia on dominant side)
* Diagnosis of Dementia
* Alcohol and/or substance abuse (in past 3 months)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2012-10; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Declarative Memory Measure - Hopkins Verbal Learning Test | Participants will be asked to complete this measure prior to the start of the intervention and again at the completion of the intervention (i.e., interval of 5 weeks between pre and post measurements).
  Individuals participating in either protocol (i.e., top-down or bottom-up) will complete the memory measure before the commencement of the treatment and again at the end of treatment.

SECONDARY OUTCOMES:
Mood Measure - Depression Anxiety Stress Scale (Lovibond & Lovibond, 1993) | Participants will be asked to complete this measure prior to the start of the intervention and again at the completion of the intervention (i.e., interval of 5 weeks between pre and post measurements).

OTHER OUTCOMES:
Functional - Multifactorial Metamemory Questionnaire (Troyer & Rich, 2011) | Participants will be asked to complete this measure prior to the start of the intervention and again at the completion of the intervention (i.e., interval of 5 weeks between pre and post measurements).

CONTACTS AND LOCATIONS:
Overall Officials: Bruno J Losier, Ph.D., Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada